CLINICAL TRIAL: NCT02529852
Title: A Phase I/II Study of Lenalidomide and Obinutuzumab With CHOP for Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0069; NCI-2015-01517 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Lymphoma
Keywords: Lymphoma; Diffuse Large B Cell Lymphoma; DLBCL; Lenalidomide; CC-5013; Revlimid; Obinutuzumab; GA101; Gazyva; Cyclophosphamide; Cytoxan; Neosar; Doxorubicin; Doxorubicin Hydrochloride; Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex; Vincristine; Prednisone
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide; obinutuzumab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide + Obinutuzumab + CHOP (Experimental): Phase I: Participants take Lenalidomide by mouth on Days 1 - 14 of each cycle. Participants receive Obinutuzumab by vein over 3 - 4 hours on Days 1, 8, and 15 of Cycle 1 and Day 1 of Cycles 2 - 6. Participants receive Cyclophosphamide by vein over about 1 hour on Day 1 of all cycles. Participants receive Doxorubicin and Vincristine by vein over about 15 minutes each on Day 1 of all cycles.
  Phase II: Participants treated at the recommended phase II dosing (RP2D) of Lenalidomide determined in the Phase Ib portion for 6 cycles of therapy. Dose of Obinutuzumab, Cyclophosphamide, Doxorubicin and Vincristine remain the same as in Phase I.
  Each study cycle is 21 days.
  Interventions: Drug: Lenalidomide; Drug: Obinutuzumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Lenalidomide — Phase I Starting Dose Level: 15 mg by mouth on Days 1 - 14 of each 21 day cycle.
  Phase II Starting Dose Level: Maximum tolerated dose from Phase I.
  Other Names: CC-5013; Revlimid
Drug: Obinutuzumab — Phase I and II: 1000 mg by vein on Days 1, 8, and 15 of Cycle 1 and Day 1 of Cycles 2 - 6.
  Other Names: GA101; Gazyva
Drug: Cyclophosphamide — Phase I and II: 750 mg/m2 vein over about 1 hour on Day 1 of all cycles.
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — Phase I and II: 50 mg/m2 by vein over about 15 minutes each on Day 1 of all cycles.
  Other Names: Doxorubicin Hydrochloride; Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex
Drug: Vincristine — Phase I and II: 1.4 mg/m2 by vein on Day 1 of all cycles.
Drug: Prednisone — Phase I and II: 100 mg by mouth daily on Days 1 - 5 of each 21 day cycle.

SUMMARY:
There are 2 parts to this study: Part 1 (dose de-escalation) and Part 2 (dose expansion).

The goal of Part 1 of this clinical research study is to find the highest tolerable dose of lenalidomide in combination with obinutuzumab and CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisone) that can be given to patients with diffuse large B cell lymphoma.

The goal of Part 2 of this clinical research study is learn if the dose of lenalidomide found in Part 1 can help to control the disease.

The safety of this drug combination will be studied in both parts.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study phase based on when you join this study. Up to 3 groups of up to 6 participants will be enrolled in Phase 1 of the study, and up to 50 participants will be enrolled in Phase 2.

If you are enrolled in Phase 1, the dose of lenalidomide you receive will depend on when you join this study. The first group of participants will receive the highest dose level of lenalidomide. Each new group will receive a lower dose of lenalidomide than the group before it, if intolerable side effects are seen. This will continue until the most tolerable dose of lenalidomide is found.

If you are enrolled in Phase 2, you will receive lenalidomide at the highest dose that was tolerated in Phase 1.

All participants will receive the same dose of CHOP and obinutuzumab.

Study Drug Administration:

Each study cycle is 21 days.

You will take lenalidomide pills by mouth on Days 1-14 of each cycle.

You will receive obinutuzumab by vein over 3-4 hours on Days 1, 8, and 15 of Cycle 1 and Day 1 of Cycles 2-6.

You will receive cyclophosphamide by vein over about 1 hour on Day 1 of all cycles.

You will receive doxorubicin and vincristine by vein over about 15 minutes each on Day 1 of all cycles.

Study Visits:

Within 3 days before Day 1 of Cycles 1-6:

* You will have a physical exam.
* Blood (about 8-9 teaspoons) will be drawn for routine tests and to check for PBMCs.

One (1) time each week during Cycle 1 and then at any time the doctor thinks it is needed, blood (about 2-3 teaspoons) will be drawn for routine tests.

At the end of Cycle 1 but before the start of Cycle 2, blood (about 6 teaspoons) will be drawn to check for PBMCs.

At the end of Cycle 3 but before the start of Cycle 4, you will have a PET/CT scan.

If you can become pregnant, blood (about 2-3 teaspoons) will be drawn for a pregnancy test 1 time before Cycle 1 and then 1 time during each cycle after that.

Length of Treatment:

You may receive lenalidomide, obinutuzumab, and CHOP therapy for up to 6 cycles. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on this study will be over after follow-up.

End-of-Treatment Visit:

Within 3-4 weeks after your last dose of study drugs:

* You will have a physical exam.
* Blood (about 8-9 teaspoons) will be drawn for routine tests and to check for PBMCs.
* You will have a PET/CT scan.
* If the doctor thinks it is needed, you will have a bone marrow biopsy to check the status of the disease.
* If the doctor thinks it is needed and the tumor is accessible, you will have a core needle biopsy to check the status of the disease. To perform a core biopsy, a sample of tissue is removed using a hollow core needle that has a cutting edge.

Follow-Up:

Every 3 months (+/- 4 weeks) during the first year after the End-of-Treatment Visit and then every 4 months (+/- 9 weeks) during the second year:

* You will have a physical exam.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You will have a PET/CT scan.

This is an investigational study. Lenalidomide is FDA approved and commercially available for the treatment of multiple myeloma (MM) and myelodysplastic syndrome (MDS). Obinutuzumab is FDA approved and commercially available for the treatment of chronic lymphocytic leukemia (CLL). CHOP is FDA approved and commercially available for the treatment of lymphoma and non-Hodgkin's lymphoma.

The combination of lenalidomide, CHOP, and obinutuzumab to treat DLBCL is considered investigational.

Up to 59 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed treatment-naïve de novo CD20+ DLBCL, regardless of cell of origin, with Stage II-IV disease, or Stage I disease if 6 cycles of chemotherapy are planned.
2. Measurable disease on cross section imaging that is at least 1.5 cm in the longest diameter and measurable in two perpendicular dimensions
3. Appropriate candidate for systemic immune-chemotherapy such as the standard RCHOP21 6 cycles as determined by the treating physician
4. Age >/=18
5. Adequate organ function (normal cardiac ejection fraction of >45%, serum bilirubin <1.5 mg/dl, AST or ALT </= 5 x ULN, and creatinine clearance > 30 mL/min (Calculated according to Cockcroft - Gault formula) unless due to lymphoma with documentation of normal function prior to onset of lymphoma. In the case of Gilberts Syndrome, or documented liver or pancreatic involvement by lymphoma, the requirement for total bilirubin is </=5.0 mg/dl
6. ANC >1000/mm3, hemoglobin >8.0, and platelets >100,000/mm3. If bone marrow is involved with lymphoma and normal marrow function prior to onset of lymphoma is documented: ANC of >750, any hemoglobin, and platelets of >50,000/mm3.
7. Performance status <3 (unless previous performance status was 0 or 1 and deterioration is due to lymphoma which treating MD expects to reverse with therapy)
8. Consent to potential need for transfusion of blood products
9. Able to give informed consent
10. Ability and willingness to comply with the requirements of the study protocol

Exclusion Criteria:

1. Prior history of low grade lymphoma with transformation to DLBCL. If a patient has a composite diagnosis of DLBCL and low grade without a prior history of lymphoma, they will not be considered ineligible.
2. Pregnant or lactating females
3. Symptomatic CNS lymphoma involvement
4. Significant comorbidity (cirrhosis, severe coronary artery disease, significant psychiatric illness, or other that may compromise the ability to safely administer the therapy at the discretion of the primary investigator)
5. HBV: Patients with positive serology for Hepatitis B defined as positivity for HBsAg or anti-HBc. Patients who are positive for anti-HBc may be considered for inclusion in the study on a case-by-case basis if they are hepatitis B viral DNA negative and are willing to undergo ongoing HBV DNA testing by real-time PCR. Patients with positive serology may be referred to a hepatologist or gastroenterologist for appropriate monitoring and management.
6. Hepatitis C (HCV): Patients with positive hepatitis C serology unless HCV RNA is confirmed negative and may be considered for inclusion in the study on a case-by-case basis.
7. Known HIV or HTLV infection
8. Previous malignancy with diagnosis or suspicion of recurrence within the past 2 years, not including non-melanoma skin cancers or in situ malignancies.
9. History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
10. Known hypersensitivity to any of the study drugs
11. Known active bacterial, viral, fungal, mycobacterial, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (related to the completion of the course of antibiotics) within 4 weeks before the start of Cycle 1
12. Major surgery (within 4 weeks prior to the start of Cycle 1), other than for diagnosis
13. Fertile men or women of childbearing potential unless 1) surgically sterile or 2) using an adequate measure of contraception such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly.
14. Effective contraception is required while receiving obinutuzumab. For women, effective contraception is required to continue for >/= 12 months after the last dose of obinutuzumab. For men, effective contraception is required to continue for 3 months after the last dose of obinutuzumab treatment.
15. Vaccination with a live vaccine a minimum of 28 days prior to the start of treatment
16. Peripheral neuropathy >/= Grade 2
17. Subjects who are unwilling to take VTE prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason R. Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Cherng HJ, Alig SK, Oki Y, Nastoupil LJ, Fayad L, Neelapu SS, Turturro F, Hagemeister F, Craig AFM, Macaulay CW, Rodriguez MA, Lee HJ, McDonnell TJ, Flowers CR, Vega F, Green MR, Feng L, Kurtz DM, Alizadeh AA, Davis RE, Westin JR. A phase 1/2 study of lenalidomide and obinutuzumab with CHOP for newly diagnosed DLBCL. Blood Adv. 2023 Apr 11;7(7):1137-1145. doi: 10.1182/bloodadvances.2022008174. PMID 36375046
- [Derived] Roschewski M, Kurtz DM, Westin JR, Lynch RC, Gopal AK, Alig SK, Sworder BJ, Cherng HJ, Kuffer C, Blair D, Brown K, Goldstein JS, Schultz A, Close S, Chabon JJ, Diehn M, Wilson WH, Alizadeh AA. Remission Assessment by Circulating Tumor DNA in Large B-Cell Lymphoma. J Clin Oncol. 2025 Dec;43(34):3652-3661. doi: 10.1200/JCO-25-01534. Epub 2025 Aug 13. PMID 40802906
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-three participants were enrolled, 6 in the phase 1b portion and 47 in the phase 2 portion. Participants started treatment between 12 November 2015 and 30 March 2017.
Pre-assignment Details: Participants were required to have adequate organ and bone marrow function. Participants were ineligible if they were pregnant or nursing women, had a prior diagnosis of low-grade lymphoma, had central nervous system involvement, active HIV infection, active Hepatitis B or C infection, or were unwilling to take aspirin for venous thrombosis prophylaxis. There was no de-escalation phase on this study.
Groups:
- Phase 1b/Phase 2: Participants were treated with Lenalidomide 15 mg orally daily on days 1 through 14 of each 21-day cycle, Obinutuzumab 1000 mg intravenously on days 1, 8, and 15 of cycle 1 and day 1 only for all additional cycles, and standard CHOP (cyclophosphamide 750 mg/m2, doxorubicin 50 mg/m2, vincristine 1.4 mg/m2 [capped at 2.0 mg], and prednisone 100 mg by mouth daily on days 1 through 5) starting on day 1 of all cycles.
Period: Overall Study
Arm/Group | Phase 1b/Phase 2
Started | 53
Phase 1b | 6
Phase 2 | 47
Completed | 51
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase1b/Phase 2: Participants were treated with Lenalidomide 15 mg orally daily on days 1 through 14 of each 21-day cycle, Obinutuzumab 1000 mg intravenously on days 1, 8, and 15 of cycle 1 and day 1 only for all additional cycles, and standard CHOP (cyclophosphamide 750 mg/m2, doxorubicin 50 mg/m2, vincristine 1.4 mg/m2 [capped at 2.0 mg], and prednisone 100 mg by mouth daily on days 1 through 5) starting on day 1 of all cycles.
Arm/Group | Phase1b/Phase 2
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 44
  More than one race | 4
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Safety of LO-CHOP
Description: Assessing the participant's characteristics and clinical outcomes after 2 cycles/42 days of LO-CHOP. The safety evaluation is defined as the lack of any grade ≥3 nonhematologic toxicity unmanageable with aggressive supportive care or toxicity, resulting in a delay of over 7 days of cycle 2.
Time Frame: up to 42 days
Population: 2 patients were inevaluable due to consent withdrawal.
Measure: Number; unit: percentage of participants
Arm/Group | Phase1b/Phase 2
Number analyzed (Participants) | 53
percentage of participants
  Grade 3 to 4 AE | 70
  DLTs | 0

2. Secondary Outcome: Overall Survival
Description: estimate overall survival
Time Frame: up to 126 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase1b/Phase 2
Number analyzed (Participants) | 53
percentage of participants | 91.3 [83.5 to 99.9]

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival
Time Frame: up to 4.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase1b/Phase 2
Number analyzed (Participants) | 53
percentage of participants | 87.4 [78.4 to 97.5]

ADVERSE EVENTS:
Time Frame: up to 4.5 years
Description: 4 patients died when already off-study, these deaths were after disease progression.
Groups:
- Phase1b/Phase2: Participants were treated with Lenalidomide 15 mg orally daily on days 1 through 14 of each 21-day cycle, Obinutuzumab 1000 mg intravenously on days 1, 8, and 15 of cycle 1 and day 1 only for all additional cycles, and standard CHOP (cyclophosphamide 750 mg/m2, doxorubicin 50 mg/m2, vincristine 1.4 mg/m2 [capped at 2.0 mg], and prednisone 100 mg by mouth daily on days 1 through 5) starting on day 1 of all cycles.
Arm/Group | Phase1b/Phase2
All-Cause Mortality (participants affected / at risk) | 4/53
Serious Adverse Events (participants affected / at risk) | 21/53
Other Adverse Events (participants affected / at risk) | 51/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase1b/Phase2 (N=53)
Neutropenia (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Fatigue (General disorders) | 7
Febrile Neutropenia (Blood and lymphatic system disorders) | 7
Infection (Infections and infestations) | 5
Pain (General disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase1b/Phase2 (N=53)
Neutropenia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Fatigue (General disorders) | 51
Febrile Neutropenia (Blood and lymphatic system disorders) | 7
Infection (Infections and infestations) | 12
Pain (General disorders) | 18
Constipation (Gastrointestinal disorders) | 45
Nausea (Gastrointestinal disorders) | 38
Anemia (Blood and lymphatic system disorders) | 33
Peripheral sensory neuropathy (Nervous system disorders) | 22
Diarrhea (Gastrointestinal disorders) | 21
Venous thromboembolism (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT02529852/Prot_SAP_000.pdf